CLINICAL TRIAL: NCT01403753
Title: Children's Familiarity With Snack Foods Changes Expectations About Fullness
Status: Completed | Type: Observational
Sponsor: University of Bristol (Other)
Responsible Party: Dr Charlotte Hardman, University of Bristol
Other Study IDs: 260608322
Record Dates: First submitted 2011-07-26; First posted 2011-07-27 (Estimated); Last update posted 2011-08-15 (Estimated); Status verified 2011-07

CONDITIONS: Children
Keywords: Obesity; Child; Dietary Habits
MeSH Terms: conditions — Obesity; Feeding Behavior

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Cross-Sectional
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (1):
- Non-clinical sample of children

SUMMARY:
The purpose of this study was to measure and quantify children's beliefs about the satiating properties (i.e. expected satiation)of snack foods. The investigators predicted that children who were especially familiar with snack foods would expect them to deliver greater satiation.

DETAILED DESCRIPTION:
Palatability is regarded as a major determinant of children's energy intake. However, few studies have considered other "non-hedonic" beliefs about foods. In adults there is emerging evidence that expectations about the satiating properties of foods are an important determinant of meal size, and that these beliefs are learned over time.

In the current study, we measured and quantified children's 'expected satiation' across energy-dense snack foods using a psychophysical technique known as method of adjustment. Participants changed a comparison-food portion (pasta and tomato sauce) to match the satiation that they expected from a snack food. We predicted that children who were especially familiar with snack foods would expect them to generate greater satiation, and that children who were unfamiliar would match expected satiation based on the physical characteristics (perceived volume) of the foods.

In our study, seventy 11- to 12-year-old children completed computerised measures of expected satiation, perceived volume, familiarity, and liking across six snack foods. Our analyses focused on the associations between these measures. This approach enabled us to establish differences in healthy behaviours that are evident across individuals.

ELIGIBILITY:
Inclusion Criteria:

* aged 11 to 12 years
* English speaking
* normal or corrected-to-normal vision

Exclusion Criteria:

* None

Ages: 11 Years to 12 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child
Study Population: Community sample
Sampling Method: Probability Sample
Enrollment: 70 (Actual)
Dates: Start 2008-08; Primary Completion 2008-12 (Actual); Study Completion 2008-12 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Jeffrey M Brunstrom, PhD, Study Director — University of Bristol
Locations (1):
- University of Bristol, Bristol, United Kingdom

REFERENCES:
- [Background] Brunstrom JM, Shakeshaft NG, Scott-Samuel NE. Measuring 'expected satiety' in a range of common foods using a method of constant stimuli. Appetite. 2008 Nov;51(3):604-14. doi: 10.1016/j.appet.2008.04.017. Epub 2008 May 1. PMID 18547677
- [Derived] Hardman CA, McCrickerd K, Brunstrom JM. Children's familiarity with snack foods changes expectations about fullness. Am J Clin Nutr. 2011 Nov;94(5):1196-201. doi: 10.3945/ajcn.111.016873. Epub 2011 Sep 14. PMID 21918214